CLINICAL TRIAL: NCT07134660
Title: Analgesic Efficacy Between Liposomal Bupivacaine and Bupivacaine Hydrochloride in Intercostal Nerve Block for Thoracic Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Thoracic Surgery Intercostal Block Trial With Liposomal vs. Hydrochloride Bupivacaine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024LY0971
Record Dates: First submitted 2025-08-03; First posted 2025-08-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain, Acute; Lung Cancer
Keywords: Postoperative Pain; Intercostal Nerve Block; Liposomal Bupivacaine
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients underwent the intervention at the end of the surgery and before regaining consciousness from anesthesia, meaning that the patients were unconscious at this time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liposomal Bupivacaine Group (Experimental): Ultrasound-guided intercostal nerve block performed at the end of surgery before emergence from anesthesia using liposomal bupivacaine 266 mg (20 mL). Patients also receive standard postoperative analgesia with IV PCA (patient-controlled analgesia) opioids and regular acetaminophen
  Interventions: Procedure: Liposomal Bupivacaine intercostal nerve block
- Bupivacaine Hydrochloride Group (Active Comparator): Ultrasound-guided intercostal nerve block performed at the end of surgery before emergence from anesthesia using 0.25% bupivacaine hydrochloride (20 mL). Patients also receive standard postoperative analgesia with IV PCA opioids and regular acetaminophen
  Interventions: Procedure: Bupivacaine Hydrochloride intercostal nerve block
- Control Group (Standard Analgesia Only) (Sham Comparator): No intercostal nerve block, just wait same time. Patients receive standard postoperative analgesia consisting of IV PCA opioids and regular acetaminophen, beginning immediately after surgery.
  Interventions: Other: Standard Postoperative Analgesia

INTERVENTIONS:
Procedure: Liposomal Bupivacaine intercostal nerve block — Ultrasound-guided intercostal nerve block with liposomal bupivacaine 266 mg (20 mL total; 4 mL per intercostal space at the incision and adjacent spaces), performed at the end of surgery before emergence from anesthesia. All patients receive standard postoperative analgesia with intravenous patient-controlled opioid analgesia.
  Arms: Liposomal Bupivacaine Group
Procedure: Bupivacaine Hydrochloride intercostal nerve block — Ultrasound-guided intercostal nerve block with 0.25% bupivacaine hydrochloride (20 mL total; 4 mL per intercostal space at the incision and adjacent spaces), performed at the end of surgery before emergence from anesthesia. All patients receive standard postoperative analgesia with intravenous patient-controlled opioid analgesia.
  Arms: Bupivacaine Hydrochloride Group
Other: Standard Postoperative Analgesia — No intercostal nerve block. Patients receive standard postoperative analgesia consisting of an intravenous patient-controlled opioid pump per institutional protocol.
  Arms: Control Group (Standard Analgesia Only)

SUMMARY:
This randomized controlled trial evaluates the analgesic effects of liposomal bupivacaine compared to bupivacaine hydrochloride in intercostal nerve block for patients undergoing thoracoscopic lung surgery. Postoperative pain remains a significant issue in thoracic procedures, often leading to complications like pneumonia or delayed recovery. The investigators hypothesize that liposomal bupivacaine, with its extended-release properties, will provide superior pain relief beyond 24 hours compared to standard bupivacaine or no block. Participants will be randomized 1:1:1 to liposomal bupivacaine group , bupivacaine hydrochloride group , or control group . Primary outcome is the area under the curve of pain scores from 25-72 hours post-surgery. Secondary outcomes include opioid consumption, recovery quality (QoR-15), and other complications.

DETAILED DESCRIPTION:
Background: Lung cancer surgery, even with minimally invasive thoracoscopy, causes significant postoperative pain in up to 62.9% of patients, potentially leading to complications and chronic pain. Intercostal nerve block is a safe alternative to epidural analgesia, but standard local anesthetics like bupivacaine provide limited duration (<8 hours). Liposomal bupivacaineoffers prolonged release up to 72 hours.

Objective: To compare the analgesic efficacy of liposomal bupivacaine versus bupivacaine hydrochloride in intercostal nerve block, assessing pain scores, opioid use, recovery quality, and complications in thoracoscopic lung surgery patients.

Design: Multicenter, randomized controlled trial with 210 participants (70 per group). Randomization with (1:1:1).

Methods: Eligible patients receive ultrasound-guided intercostal block post-surgery: Liposomal bupivacaine (20 mL, 266 mg), bupivacaine HCl (20 mL, 0.25%), or control (IV PCA only). Follow-up includes pain scores, opioid consumption, QoR-15, and adverse events up to 72 hours.

Expected Outcomes: Liposomal bupivacaine expected to reduce pain AUC by >10% vs. bupivacaine and >15% vs. control from 25-72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective unilateral thoracoscopic (VATS) lung surgery
* Age 18 to 80 years
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Contraindication to local anesthetics (infection at puncture site, allergy to local anesthetics, coagulopathy or other bleeding risk)
* Sensory abnormalities in the planned chest-wall surgical area
* Hepatic dysfunction (ALT > 50 U/L, AST > 40 U/L, or total bilirubin ≥ 19 μmol/L) or renal dysfunction (serum creatinine > 112 μmol/L, BUN > 7.1 mmol/L, or dialysis within 28 days before surgery)
* Pregnancy, breastfeeding, women of childbearing potential not using adequate contraception, or planning pregnancy during the study period
* Preoperative opioid use, history of chronic pain, or history of opioid abuse
* Refusal to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain score area under the curve (AUC) from 25 to 72 hours postoperatively | 25 to 72 hours after the end of surgery
  Area under the curve of postoperative pain intensity measured on the VRS. AUC is computed over the 25-72 h interval. Postoperative pain intensity assessed using the Verbal Response Scale (VRS), the score ranges from 0 to 10, with a total of 11 numbers corresponding to different pain levels: 0 indicates no pain; 1-3 indicates mild pain (tolerable and does not affect sleep); 4-6 indicates moderate pain (significant, affects sleep, and requires medication for relief); and 7-10 indicates severe pain (intense, intolerable, and severely affects life).

SECONDARY OUTCOMES:
Pain score at PACU discharge and postoperative intervals | At PACU discharge, and 6, 12, 24, 48, and 72 hours postoperatively
  Pain intensity assessed using the VRS in the post-anesthesia care unit (PACU) and at 6, 12, 24, 48, and 72 hours after surgery. Postoperative pain intensity assessed using the Verbal Response Scale (VRS), the score ranges from 0 to 10, with a total of 11 numbers corresponding to different pain levels: 0 indicates no pain; 1-3 indicates mild pain (tolerable and does not affect sleep); 4-6 indicates moderate pain (significant, affects sleep, and requires medication for relief); and 7-10 indicates severe pain (intense, intolerable, and severely affects life).Rescue analgesia is provided if VRS >4.
Cumulative opioid consumption | From the end of surgery to 48 hours after surgery
  Total postoperative opioid use converted to morphine milligram equivalents.

OTHER OUTCOMES:
Duration of chest wall analgesia | From intervention (end of surgery) up to 7 days
  Time from performance of the intercostal nerve block (end of surgery) to return of chest-wall sensation, as determined by cold and pinprick testing at predefined chest-wall sites.
Quality of Recovery (QoR-15) score | 24, 48, and 72 hours after surgery
  Measured by the QoR-15 questionnaire (15 items, total score 0-150; higher scores indicate better recovery).
Incidence of postoperative nausea and vomiting | 24, 48, and 72 hours postoperatively
  Number of patients of nausea or vomiting recorded at 24, 48, and 72 hours after surgery.
Incidence of postoperative pulmonary complications | From intervention (end of surgery) up to 7 days
  Occurrence of postoperative pulmonary complications-including pneumonia, atelectasis, acute respiratory distress syndrome (ARDS), and aspiration-defined by CDC and Berlin criteria.
Length of hospital stay | From intervention (end of surgery) up to 7 days
  Time from end of surgery to discharge, measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Y Lv, PhD, Study Director — Shanghai Pulmonary Hospital, Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Wang L, Wei S, Xin Y, Chang R, Liu H, Yang Y, Song J, Lv X. Comparison of liposomal bupivacaine and bupivacaine hydrochloride intercostal nerve blocks for postoperative analgesia after thoracic surgery: a multicenter, randomized, three arms trial protocol. Ann Med. 2026 Dec;58(1):2612384. doi: 10.1080/07853890.2025.2612384. Epub 2026 Jan 20. PMID 41560407
- [Derived] Yu J, Wei S, Ling D, Xin Y, Liu H, Yang Y, Li X, Xiang Z, Liu J. Effective Dose of Oliceridine for Inhibiting Hemodynamic Elevation Induced by Tracheal Intubation: An Up-and-Down Sequential Trial. Drug Des Devel Ther. 2025 Dec 26;19:11767-11778. doi: 10.2147/DDDT.S567868. eCollection 2025. PMID 41477178